CLINICAL TRIAL: NCT06457893
Title: THE EFFECT OF THE EDUCATION PROGRAM BASED ON THE HEALTH BELIEF MODEL ON THE PHYSICAL ACTIVITY BELIEFS AND BEHAVIOR OF FIRST YEAR STUDENTS OF THE FACULTY OF NURSING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, AYLA AYKAC KOCAK, PHD STUDENT, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: E-76261397-050.99-167339
Record Dates: First submitted 2024-06-09; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: THE HEALTH BELIEF MODEL ON THE PHYSICAL ACTIVITY BELIEFS
Keywords: Youth; Exercise Training; Exercise; Physical Inactivity; Physical Activity
MeSH Terms: conditions — Motor Activity; Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: Structured education and physical activity.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Experimental): The study includes with a total of 121 students, 60 in the experimental group and 61 in the control group. No intervention will be made to the students in the control group
  Interventions: Other: The health belief model-based exercise training program and health belief model-based education
- Experimental Group (Experimental): The study includes with a total of 121 students, 60 in the experimental group and 61 in the control group. The health belief model-based exercise training program will implement with the students in the experimental group for 5 weeks and follow-ups will be made at the 3rd and 6th months.
  Interventions: Other: The health belief model-based exercise training program and health belief model-based education

INTERVENTIONS:
Other: The health belief model-based exercise training program and health belief model-based education — The health belief model-based exercise training program and education program will implement with the students in the experimental group for 5 weeks and follow-ups will be made at the 3rd and 6th months.

SUMMARY:
The aim of the study is to examine the effect of the Health Belief Model-Based Education Program on the Physical Activity Beliefs and Behaviors of First Year Students of the Faculty of Nursing using a randomized controlled experimental research method.

DETAILED DESCRIPTION:
The research was conducted in a randomized controlled manner between December 2022 and October 2023, among first-year students of the faculty of nursing who wanted to participate in an education program based on the health belief model. The study was completed with a total of 121 students, 60 in the experimental group and 61 in the control group. The health belief model-based exercise training program was implemented with the students in the experimental group for 5 weeks and follow-ups were made at the 3rd and 6th months. No intervention was made to the students in the control group. Experimental and control group data were collected with the Student Personal Information Form, Exercise Health Belief Model Scale and International Physical Activity Short Survey Form. Data were evaluated with descriptive statistics, Mann Whitney-U, Chi-square, Independent Sample T Test, Paired Sample Test and ANOVA analysis.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years of age
* No language barrier in communication.
* Not having any disease or illness (arrhythmia, heart disease, bronchitis, chronic herniated disc pain, chronic neck herniated pain) that would prevent participation in the study.
* Not having received structured training for physical activity.

Exclusion Criteria:

* Foreign students
* Students who fill out any of the forms related to the study incompletely (experiment, control)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2022-12-19 (Actual); Primary Completion 2023-01-19 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Health Belief Model Scale Scores | 6 months
  Checking change in the exercise health belief model scale scores of the control group students .

CONTACTS AND LOCATIONS:
Overall Officials: AYLA AYKAC KOCAK, Principal Investigator — Aydin Adnan Menderes University
Locations (1):
- Aydin Adnan Menderes University, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
IPD Plan Description:
  The data sets generated during and/or analyzed during the current study are available from the corresponding author on reasonable request.
  IPD Sharing Access Criteria:
  Relevance to the topic of the study and approval of all co-authors within 1 month of receiving the request.
  IPD Sharing Time Frame:
  6 months after publication
  IPD Sharing Supporting Information Type:
  Clinical Study Report (CSR)